CLINICAL TRIAL: NCT07199088
Title: Comparative Efficacy and Safety of Acetazolamide Versus Metolazone as an Adjunct to Standard Therapy in Patients With Acute Decompensated Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dr. Matiullah Azmoon, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 772
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Decompensated Heart Failure; Heart Failure, Diastolic; Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure, Systolic | interventions — Acetazolamide; Metolazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide + Standard Therapy (Experimental): Participants in this group will receive acetazolamide (500 mg/day) as an adjunct to standard heart failure therapy, which includes intravenous loop diuretics (Furosemide 80 mg/day). This group aims to assess the efficacy and safety of acetazolamide in improving decongestion in patients with acute decompensated heart failure.
  Interventions: Other: Acetazolamide
- Metolazone Group (Active Comparator): Participants in this group will receive metolazone (5 mg/day) as an adjunct to standard heart failure therapy, including intravenous loop diuretics (Furosemide 80 mg/day). This group serves as a comparison to the acetazolamide group, evaluating the efficacy and safety of metolazone in improving decongestion in patients with acute decompensated heart failure.
  Interventions: Other: Metolazone

INTERVENTIONS:
Other: Acetazolamide — A carbonic anhydrase inhibitor, 500 mg orally once a day as an adjunct to loop diuretics for enhancing diuresis and improving decongestion in ADHF patients.
  Arms: Acetazolamide + Standard Therapy
Other: Metolazone — A thiazide-like diuretic, 5 mg orally once a day as an adjunct to loop diuretics for enhancing diuresis and improving decongestion in ADHF patients.
  Arms: Metolazone Group

SUMMARY:
This clinical trial aims to compare the efficacy and safety of acetazolamide versus metolazone as adjunctive treatments to standard therapy in patients with acute decompensated heart failure (ADHF). ADHF is a life-threatening condition, and current treatments often involve loop diuretics to alleviate volume overload. This study will assess the added benefit of acetazolamide and metolazone in improving decongestion, reducing hospital stays, and preventing complications such as renal dysfunction or electrolyte imbalances. Participants will be randomized to receive either acetazolamide or metolazone in addition to standard diuretic therapy. The trial will evaluate primary outcomes including successful decongestion, in-hospital mortality, and length of hospital stay, with secondary outcomes focusing on renal function, electrolyte disturbances, and overall safety. The study is conducted at Bahawal Victoria Hospital, Bahawalpur, and aims to provide valuable insights into the management of ADHF, especially in the Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Diagnosed with Acute Decompensated Heart Failure (ADHF), with either preserved or reduced ejection fraction (EF).
* At least one clinical sign of volume overload, such as:
* Pleural effusion (confirmed by chest X-ray or ultrasound).
* Oedema or ascites (verified by abdominal ultrasonography).
* Plasma NT-proBNP level > 1000 pg/mL or BNP level > 250 ng/mL at screening.
* Receiving at least 40 mg of furosemide as oral maintenance therapy for at least one month prior to the study initiation.

Exclusion Criteria:

* Previous use of acetazolamide or metolazone prior to the study period.
* Known hypersensitivity or allergies to the study drugs (acetazolamide or metolazone) or their components.
* Patients with electrolyte disturbances, especially hypokalemia.
* End-stage renal disease requiring dialysis or GFR < 20 mL/min/1.73 m².
* Pregnant or breastfeeding women.
* Severe hypotension (systolic blood pressure < 90 mmHg) or other significant comorbidities like congenital cardiac illness requiring surgery.
* Patients requiring renal replacement therapy during the hospitalization.
* History of significant electrolyte imbalances or acid-base disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-10-11 (Estimated); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Successful Decongestion | 72 hours after randomization (following 3 days of treatment with the assigned adjunct therapy).
  This outcome measure assesses the resolution of clinical signs and symptoms of acute decompensated heart failure (ADHF), specifically the absence of orthopnea, reduced jugular venous distention (JVD) to <8 cm H2O, and minimal or no peripheral edema. Successful decongestion is considered when these signs are resolved within 72 hours of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Quaid e Azam Medical College , bahawalpur, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided